CLINICAL TRIAL: NCT03668236
Title: The Conservative vs. Liberal Approach to Fluid Therapy of Septic Shock in Intensive Care Trial
Acronym: CLASSIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anders Perner, MD, PhD (Other)
Collaborators: Rigshospitalet, Denmark (Other); Centre for Research in Intensive Care (CRIC) (Other); Scandinavian Critical Care Trials Group (Other)
Responsible Party: Sponsor-Investigator, Anders Perner, MD, PhD, MD, PhD, Senior staff specialist , Professor in Intensive Care, Scandinavian Critical Care Trials Group
Organization: Scandinavian Critical Care Trials Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RH-ITA-007
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Septic Shock
Keywords: Fluid resuscitation; Critical care; Intensive care; Crystalloid; IV fluid therapy
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor- and analyst-blinded trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid restriction group (Experimental): No IV fluids unless one of the extenuating circumstances occur; then, IV fluid may be given in measured amounts:
  1. In case of severe hypoperfusion or severe circulatory impairment defined by either:
     * Lactate≥4 mmol/L
     * MAP<50 mmHg (with or without vasopressor/inotrope)
     * Mottling beyond the kneecap (mottling score >2) OR
     * Urinary output<0.1 mL/kg bodyweight/h, but only in the first 2hrs after randomisation
     A bolus of 250-500 ml of IV crystalloid solution may be given followed by re-evaluation
  2. In case of overt fluid losses (e.g. vomiting, large aspirates,…) IV fluid may be given to correct for the loss, but not above the volume lost.
  3. In case the oral/enteral route for water or electrolyte solutions is contraindicated or has failed, IV fluids may be given to:
     * Correct dehydration or electrolyte deficiencies
     * Ensure a total fluid input of 1L per 24hrs
  IV fluids may be given as carrier for medication, but the volume should be reduced to the lowest possible
  Interventions: Drug: Isotonic crystalloids
- Standard-care (Active Comparator): There will be no upper limit for the use of either IV or oral/enteral fluids. In particular:
  1. IV fluids should be given in the case of hypoperfusion or circulatory impairment and should be continued as long as hemodynamic variables improve including static or dynamic variable(s) as chosen by the clinicians. These criteria are based on the Surviving Sepsis Campaign guideline.
  2. IV fluids should be given as maintenance if the ICU has a protocol recommending maintenance fluid
  3. IV fluids should be given to substitute expected or observed loss, dehydration or electrolyte derangements
  Interventions: Drug: Isotonic crystalloids

INTERVENTIONS:
Drug: Isotonic crystalloids — Types of fluid to be used in both intervention groups:
  * IV fluids given for circulatory impairment: Only isotonic crystalloids are to be used as per the Scandinavian guideline for fluid resuscitation
  * Fluids given to substitute overt loss: Isotonic crystalloids are to be used. If large amounts of ascites are tapped, then human albumin may be used
  * Fluids used for dehydration: Water or isotonic glucose should be used
  * Fluids used for electrolyte disturbances: Fluids should be chosen to substitute the specific deficiency, including water in the case of severe hypernatremia
  * Blood products are only to be used on specific indications including severe bleeding, severe anaemia and prophylactic in case of severe coagulopathy

SUMMARY:
The purpose of this trial is to assess patient important benefits and harms of IV fluid restriction vs. standard care fluid therapy in patients with septic shock.

DETAILED DESCRIPTION:
BACKGROUND:

Septic shock is common, often lethal, costly, and associated with prolonged suffering among survivors and relatives. Traditionally, intravenous (IV) fluids are used to optimise the circulation, and the use of higher volumes is recommended by international guidelines. There is, however, no high-quality evidence to support this. In contrast, data from cohort studies, small trials and systematic reviews in sepsis and large trials in other settings and patient groups suggest potential benefits from restriction of IV fluids in patients with septic shock.

OBJECTIVES:

The aim of the CLASSIC trial is to assess the benefits and harms of IV fluid restriction vs. standard care on patient-important outcome measures in adult intensive care unit (ICU) patients with septic shock.

DESIGN:

CLASSIC is an international, multicentre, parallel-grouped, open-labelled, centrally randomised, stratified, outcome assessor- and analyst-blinded trial.

POPULATION:

Adult ICU patients who have septic shock and have received at least 1 L of IV fluid in the last 24-hours.

EXPERIMENTAL INTERVENTION:

In the IV fluid restriction group no IV fluids should be given in the ICU unless extenuating circumstances occur, including signs of severe hypoperfusion, overt fluid loss or a failing GI tract with a total fluid input of less than 1 L per day. In these circumstances, IV fluid may be given in measured amounts.

CONTROL INTERVENTION:

In the standard care group there will be no upper limit for the use of IV fluids.

OUTCOMES:

The primary outcome is 90-day mortality; secondary outcomes are serious adverse events in the ICU (ischemic events or severe acute kidney injury); serious adverse reactions in the ICU; days alive without life support at day 90; days alive and out of hospital at day 90 and mortality, health-related quality of life and cognitive function at 1-year.

TRIAL SIZE:

A total of 1554 participants will be randomised to allow the detection of a 15% relative risk reduction (7% absolute) in the restrictive vs. standard care group in 90-day mortality with a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria must be fulfilled:

* Aged 18 years or above
* Admitted to the ICU or plan to be admitted to the ICU regardless of trial participation
* Septic shock defined according to the Sepsis-3 criteria:

  * Suspected or confirmed site of infection or positive blood culture AND
  * Ongoing infusion of vasopressor/inotrope agent to maintain a mean arterial blood pressure of 65 mmHg or above AND
  * Lactate of 2 mmol/L or above in any plasma sample performed within the last 3-hours
* Have received at least 1 L of IV fluid (crystalloids, colloids or blood products) in the last 24-hours prior to screening.

Exclusion Criteria:

Patients who fulfil any of the following criteria will be excluded:

* Septic shock for more than 12 hours at the time of screening as these patients are no longer early in their course
* Life-threatening bleeding as these patients need specific fluid/blood product strategies
* Acute burn injury of more than 10% of the body surface area as these patients need a specific fluid strategy
* Known pregnancy
* Consent not obtainable as per the model approved for the specific site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1554 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tine Sylvest Meyhoff, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (31):
- University Hospital Brussels (UZB), Brussels, Belgium
- Medical Intensive Care Unit, Fakultni Nemocnice, Pilsen, Czechia
- Denmark (11):
  - Dept. of Anaesthesia and Intensive Care, Aalborg University Hospital, Denmark., Aalborg
  - Dept of Intensive Care,Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Dept. of Anaesthesia and Intensive Care, Bispebjerg Hospital, Copenhagen
  - Dept. of Anaesthesia and Intensive Care, Herning Hospital, Herning
  - Dept. of Intensive Care, Hillerød Hospital, Hillerød
  - Dept. of Anaesthesia and Intensive Care, Holbæk Hospital, Holbæk
  - Dept. of Anaesthesia and Intensive Care, Lillebaelt Hospital, Kolding
  - Dept. of Anaesthesia and Intensive Care, Zealand University Hospital Køge, Køge
  - Dept. of Anaesthesia and Intensive Care, Randers Hospital, Randers
  - Dept. of Anaesthesia and Intensive Care, Zealand University Hospital Roskilde, Roskilde
  - Dept. of Anaesthesia and Intensive Care, Viborg Hospital, Viborg
- Italy (4):
  - Humanitas research hospital Bergamo, Bergamo, Milan
  - Dept. of Intensive Care, Humanitas Research Hospital Castelanza, Castellanza, Milan
  - Dept. of Intensive Care, Ancona Hospital, Ancona
  - Dept. of Intensive Care, Humanitas Research Hospital, Milan
- Norway (4):
  - Dept. of intensive care, Østfold, Kalnes, Grålum
  - Dept. of intensive Care, Innlandet Hamar, Hamar
  - Dept. of Intensive Care, Oslo University Hospital, Oslo
  - Dept. of Intensive Care Medicine, Stavanger, Stavanger
- Sweden (7):
  - Dept. of Intensive Care Medicine, St Göran, Gothenburg
  - Dept. of intensive care, Huddinge, Huddinge
  - MIMA Medicinsk intermediärvårdsavdelning, Huddinge
  - Dept. of Intensive Care, Solna, Solna
  - Medical ICU, Karolinska, Södersjukhuset, Stockholm
  - Södersjukhuset, Stockholm
  - Dept. of Intensive Care Medicine Sundsvall Hospital, Sundsvall
- Switzerland (2):
  - Dept. of intensive care, Basel, Basel
  - Dept. of Intensive Care, University Hospital Bern, Bern
- Dept. of Intensive Care Unit, Guy's and St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hjortrup PB, Haase N, Bundgaard H, Thomsen SL, Winding R, Pettila V, Aaen A, Lodahl D, Berthelsen RE, Christensen H, Madsen MB, Winkel P, Wetterslev J, Perner A; CLASSIC Trial Group; Scandinavian Critical Care Trials Group. Restricting volumes of resuscitation fluid in adults with septic shock after initial management: the CLASSIC randomised, parallel-group, multicentre feasibility trial. Intensive Care Med. 2016 Nov;42(11):1695-1705. doi: 10.1007/s00134-016-4500-7. Epub 2016 Sep 30. PMID 27686349
- [Background] Meyhoff TS, Hjortrup PB, Wetterslev J, Sivapalan P, Laake JH, Cronhjort M, Jakob SM, Cecconi M, Nalos M, Ostermann M, Malbrain M, Pettila V, Moller MH, Kjaer MN, Lange T, Overgaard-Steensen C, Brand BA, Winther-Olesen M, White JO, Quist L, Westergaard B, Jonsson AB, Hjortso CJS, Meier N, Jensen TS, Engstrom J, Nebrich L, Andersen-Ranberg NC, Jensen JV, Joseph NA, Poulsen LM, Herlov LS, Solling CG, Pedersen SK, Knudsen KK, Straarup TS, Vang ML, Bundgaard H, Rasmussen BS, Aagaard SR, Hildebrandt T, Russell L, Bestle MH, Schonemann-Lund M, Brochner AC, Elvander CF, Hoffmann SKL, Rasmussen ML, Martin YK, Friberg FF, Seter H, Aslam TN, Adnoy S, Seidel P, Strand K, Johnstad B, Joelsson-Alm E, Christensen J, Ahlstedt C, Pfortmueller CA, Siegemund M, Greco M, Radej J, Kriz M, Gould DW, Rowan KM, Mouncey PR, Perner A; CLASSIC Trial Group. Restriction of Intravenous Fluid in ICU Patients with Septic Shock. N Engl J Med. 2022 Jun 30;386(26):2459-2470. doi: 10.1056/NEJMoa2202707. Epub 2022 Jun 17. PMID 35709019
- [Background] Meyhoff TS, Hjortrup PB, Moller MH, Wetterslev J, Lange T, Kjaer MN, Jonsson AB, Hjortso CJS, Cronhjort M, Laake JH, Jakob SM, Nalos M, Pettila V, van der Horst I, Ostermann M, Mouncey P, Rowan K, Cecconi M, Ferrer R, Malbrain MLNG, Ahlstedt C, Hoffmann S, Bestle MH, Nebrich L, Russell L, Vang M, Rasmussen ML, Solling C, Rasmussen BS, Brochner AC, Perner A. Conservative vs liberal fluid therapy in septic shock (CLASSIC) trial-Protocol and statistical analysis plan. Acta Anaesthesiol Scand. 2019 Oct;63(9):1262-1271. doi: 10.1111/aas.13434. Epub 2019 Jul 24. PMID 31276193
- [Derived] Sivapalan P, Kaas-Hansen BS, Meyhoff TS, Hjortrup PB, Kjaer MN, Laake JH, Cronhjort M, Jakob SM, Cecconi M, Nalos M, Ostermann M, Malbrain MLNG, Moller MH, Perner A, Granholm A. Effects of IV Fluid Restriction According to Standard Fluid Treatment Intensity Across Conservative Versus Liberal Approach to Fluid Therapy of Septic Shock in Intensive Care (CLASSIC) Trial Sites. Crit Care Med. 2025 Aug 1;53(8):e1590-e1600. doi: 10.1097/CCM.0000000000006679. Epub 2025 Apr 24. PMID 40272936
- [Derived] Sivapalan P, Kaas-Hansen BS, Meyhoff TS, Hjortrup PB, Kjaer MN, Laake JH, Cronhjort M, Jakob SM, Cecconi M, Nalos M, Ostermann M, Malbrain MLNG, Moller MH, Perner A, Granholm A. Effects of IV fluid restriction according to site-specific intensity of standard fluid treatment-protocol. Acta Anaesthesiol Scand. 2024 Aug;68(7):975-982. doi: 10.1111/aas.14423. Epub 2024 Apr 4. PMID 38576165
- [Derived] Kjaer MN, Meyhoff TS, Sivapalan P, Granholm A, Hjortrup PB, Madsen MB, Moller MH, Egerod I, Wetterslev J, Lange T, Cronhjort M, Laake JH, Jakob SM, Nalos M, Ostermann M, Gould D, Cecconi M, Malbrain MLNG, Ahlstedt C, Kiel LB, Bestle MH, Nebrich L, Hildebrandt T, Russell L, Vang M, Rasmussen ML, Solling C, Brochner AC, Krag M, Pfortmueller C, Kriz M, Siegemund M, Albano G, Aagaard SR, Bundgaard H, Crone V, Wichmann S, Johnstad B, Martin YK, Seidel P, Martensson J, Hollenberg J, Wistrand M, Donati A, Barbara E, Karvunidis T, Hollinger A, Carsetti A, Lumlertgul N, Joelsson-Alm E, Lambiris N, Aslam TN, Friberg FF, Vesterlund GK, Mortensen CB, Vestergaard SR, Caspersen SF, Jensen DB, Borup M, Rasmussen BS, Perner A. Long-term effects of restriction of intravenous fluid in adult ICU patients with septic shock. Intensive Care Med. 2023 Jul;49(7):820-830. doi: 10.1007/s00134-023-07114-8. Epub 2023 Jun 18. PMID 37330928
- [Derived] Meyhoff TS, Moller MH, Hjortrup PB, Cronhjort M, Perner A, Wetterslev J. Lower vs Higher Fluid Volumes During Initial Management of Sepsis: A Systematic Review With Meta-Analysis and Trial Sequential Analysis. Chest. 2020 Jun;157(6):1478-1496. doi: 10.1016/j.chest.2019.11.050. Epub 2020 Jan 23. PMID 31982391
- [Derived] Kjaer MN, Meyhoff TS, Madsen MB, Hjortrup PB, Moller MH, Egerod I, Wetterslev J, Lange T, Cronhjort M, Laake JH, Jakob SM, Nalos M, Pettila V, van der Horst ICC, Ostermann M, Mouncey P, Cecconi M, Ferrer R, Malbrain MLNG, Ahlstedt C, Hoffmann S, Bestle MH, Gyldensted L, Nebrich L, Russell L, Vang M, Solling C, Brochner AC, Rasmussen BS, Perner A. Long-term patient-important outcomes after septic shock: A protocol for 1-year follow-up of the CLASSIC trial. Acta Anaesthesiol Scand. 2020 Mar;64(3):410-416. doi: 10.1111/aas.13519. Epub 2019 Dec 26. PMID 31828753
- See also: Official study website — http://www.cric.nu/classic/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were excluded from the trial prior to group assignment.
Groups:
- Fluid Restriction Group: No IV fluids unless one of the extenuating circumstances occurred (additional details in protocol section)
- Standard-care: No upper limit for IV fluids (additional details in protocol section).
Period: Randomization
Arm/Group | Fluid Restriction Group | Standard-care
Started | 770 | 784
Completed | 770 | 784
Not Completed | 0 | 0
Period: 90-day Follow-up
Arm/Group | Fluid Restriction Group | Standard-care
Started | 770 | 784
Completed | 764 | 781
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 3 | 1
Period: Baseline Characteristics
Arm/Group | Fluid Restriction Group | Standard-care
Started | 764 | 781
Completed | 755 | 776
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 9 | 5
Period: 1-year Follow-up
Arm/Group | Fluid Restriction Group | Standard-care
Started | 767 | 782
Completed | 750 | 767
Not Completed | 17 | 15
Not completed — Withdrawal by Subject | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluid Restriction Group | Standard-care | Total
Number analyzed (Participants) | 755 | 776 | 1531
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [62 to 77] | 70 [60 to 77] | 70 [61 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303 | 324 | 627
  Male | 452 | 452 | 904
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 755 | 776 | 1531
Volume of intravenous fluid 24 hr before randomization [Median (Inter-Quartile Range); unit: ml] | 3200 [2000 to 4700] | 3000 [2000 to 4842] | 3068 [2000 to 4740]

OUTCOME MEASURES:

1. Primary Outcome: 90-day Mortality
Description: Al cause mortality at 90 days
Time Frame: Day 90 after randomisation
Population: Primary outcome data were missing from six patients in the restrictive-fluid group and three in the standard-fluid group.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 764 | 781
Participants | 323 | 329

2. Secondary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs) in the ICU
Description: SAEs were defined as ischaemic events (cerebral, cardiac, intestinal or limb ischaemia) or as a new episode of severe acute kidney injury (modified KDIGO-3)
Time Frame: Until ICU discharge, maximum 90 days
Population: All secondary outcome data were missing for 23 patients (15 patients in the restrictive-fluid group and 8 in the standard-fluid group). In the analysis of SAEs in the ICU, additional 9 patients (5 in the restrictive-fluid group and 4 in the standard-fluid group) had missing data for severe acute kidney injury. One of the 5 patients in the restrictive-fluid group had another SAE; thus only 8 patients had missing data in the composite outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 751 | 772
Participants | 221 | 238

3. Secondary Outcome: Number of Participants With One or More Serious Adverse Reactions (SARs) to IV Crystalloids in the ICU.
Description: The pre-specified SARs to IV crystalloids were: Generalized tonic-clonic seizures, anaphylactic reactions, central pontine myelinolysis, severe hypernatremia, severe hyperchloremic acidosis, and severe metabolic alkalosis. Data on the outcome measures, including SARs, were obtained from patient medical records by the trial investigators or their delegates.
Time Frame: Until ICU discharge, maximum 90 days
Population: All secondary outcome data were missing for 23 patients (15 patients in the restrictive-fluid group and 8 in the standard-fluid group).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 755 | 776
Participants | 31 | 32

4. Secondary Outcome: Days Alive at Day 90 Without Life Support (Vasopressor / Inotropic Support, Invasive Mechanical Ventilation or Renal Replacement Therapy)
Time Frame: Until ICU discharge, maximum 90 days
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 755 | 776
days | 77 [1 to 87] | 77 [1 to 87]

5. Secondary Outcome: Days Alive and Out of Hospital at Day 90
Time Frame: Day 90 after randomisation
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 755 | 776
days | 21 [0 to 69] | 33 [0 to 70]

6. Secondary Outcome: All-cause Mortality at 1-year After Randomisation
Time Frame: 1-year after randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 750 | 767
Participants | 385 | 383

7. Secondary Outcome: Health-related Quality of Life 1 Year After Randomisation
Description: Measured using the EuroQoL EQ-5D-5L questionnaire (comprising 5 questions with a score from 1 to 5 each and a visual analogue scale from 0 to 100). Participants who have died will be assigned the lowest possible scores.
Time Frame: 1 year after randomisation
Population: In total, 46 patients in the restrictive group and 55 in the standard group had missing data (either completely missing or partially missing) for EQ-5D-5L index values.
Measure: Median (Inter-Quartile Range); unit: EQ-5D-5L index values
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 704 | 712
EQ-5D-5L index values | 0 [0 to 0.82] | 0 [0 to 0.81]

8. Secondary Outcome: Cognitive Function 1-year After Randomisation
Description: Assessed by the Montreal Cognitive Assessment (MoCa) MINI score validated for telephone use. Mini MoCA consists of 4 cognitive dimensions: attention (immediate recall of 5 words), executive functions and language (1-min verbal fluency), orientation (6 items on date and geographic orientation), and memory (delayed recall and recognition of 5 previously learned words). The total score ranges from 0 to 30, with lower values indicating worse cognitive function. To correct for any educational effect on the cognitive test, 1 point is added for participants with 12 years of education or less (scores were truncated at the maximum upper value of 30 points) Participants who had died were assigned the value 0.
Time Frame: 1-year after randomisation
Population: In total, 82 patients in the restrictive group and 98 in the standard group had missing data (either completely missing or partially missing) for Mini MOCA.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Fluid Restriction Group | Standard-care
Number analyzed (Participants) | 668 | 669
Units on a scale | 0 [0 to 22] | 0 [0 to 22]

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed until ICU discharge, maximum 90 days. All-cause mortality was assessed during ICU stay and continued following discharge from the ICU to 90 days and 1-year from randomization, respectively. "At risk" population for mortality at 90 days was 764 in the restrictive group and 781 in the standard group. At 1-year, the "at risk" population for mortality was 750 patients in the fluid restriction group, and 767 in the standard group, due to withdrawn consent.
Description: Serious adverse events (SAEs), excluding mortality, was a secondary outcome. All secondary outcome data were missing for 15 patients in the restrictive group and 8 in the standard group. For SAEs, additional 5 patients in the restrictive group and 4 in the standard group had missing data for severe acute kidney injury. One of the 5 patients in the restrictive group had another SAE. For mortality, data were missing from 6 patients in the restrictive group and 3 in the standard group.
Arm/Group | Fluid Restriction Group | Standard-care
All-Cause Mortality (participants affected / at risk) | 385/764 | 383/781
Serious Adverse Events (participants affected / at risk) | 221/755 | 238/776
Other Adverse Events (participants affected / at risk) | 0/755 | 0/776
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fluid Restriction Group (N=755) | Standard-care (N=776)
Cerebral ischemia (General disorders) | 17 | 18
Myocardial ischemia (General disorders) | 16 | 6
Intestinal ischemia (General disorders) | 41 | 44
Limb ischemia (General disorders) | 18 | 18
Severe acute kidney injury (General disorders) | 173/750 | 189/772

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03668236/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03668236/SAP_001.pdf